CLINICAL TRIAL: NCT03286075
Title: Impact of Transcranial Direct Current Stimulation of the Dorsolateral Prefrontal Cortex on Emotional Processing in Healthy Subjects.
Brief Title: Impact of tDCS on Emotional Processing in Healthy Subjects.
Acronym: EmoStimH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The department in charge of this research is no longer able to follow this project. Only two inclusions this study is close
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 2016-A01258-43
Record Dates: First submitted 2017-09-12; First posted 2017-09-18 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Transcranial Direct Current Stimulation
Keywords: DLPFC, tDCS, emotional processing

STUDY DESIGN:
Intervention Model Description: 3 arms will take part in the study: Anode tDCS Cathode tDCS Placebo tDCS These 3 types of tDCS stimulation will enable us to study the different modulations possible for the DLPFC and the impact on all the variables previously mentioned
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anode tDCS (Experimental): The subjects in this arm will undertake a unique session of tDCS on the DLPFC (anode on the left DLPF).
  Subjects will receive a 30-minutes session of 2mA tDCS. Facial emotion recognition task and attentional and working memory tasks with measurement of eye-tracking, heart rate, respiratory frequency and skin conductance will be conducted before and after the session.
  Interventions: Device: tDCS Anode session
- Cathode tDCS (Experimental): The subjects in this arm will undertake a unique session of tDCS on the DLPFC (cathode on the left DLPF).
  Subjects will receive a 30-minutes session of 2mA tDCS. Facial emotion recognition task and attentional and working memory tasks with measurement of eye-tracking, heart rate, respiratory frequency and skin conductance will be conducted before and after the session.
  Interventions: Device: tDCS Cathode session
- Placebo tDCS (Placebo Comparator): The subjects in this arm will undertake a unique session of tDCS on the DLPFC (placebo).
  Subjects will receive a 30-minutes SHAM session of tDCS.
  Interventions: Device: tDCS Placebo session

INTERVENTIONS:
Device: tDCS Anode session — The aim of this unique anode tDCS session is to study the possibility of enhancing emotional processing, attentional resources and physiological responses in healthy subjects.
  The arm will be compared to the other 2, enabling us to compare different tDCS stimulation modes.
  Stimulation will be performed using a tDCS stimulator (Neuroconn or Neuroelectric tDCS stimulator) with two 7×5 cm (35 cm2) sponge electrodes soaked in a saline solution (0.9% NaCl) Anode will be placed over the left dorsolateral prefrontal cortex (F3 according to the international EEG system) and cathode over the right dorsolateral prefrontal cortex (F4 according to the international EEG system).
  Arms: Anode tDCS
Device: tDCS Cathode session — The aim of this unique cathode tDCS session is to study the possibility of inhibiting or altering emotional processing, attentional resources and physiological responses in healthy subjects.
  This arm will be compared to the other 2, enabling us to compare different tDCS stimulation modes.
  Stimulation will be performed using a tDCS stimulator (Neuroconn or Neuroelectric tDCS stimulator) with two 7×5 cm (35 cm2) sponge electrodes soaked in a saline solution (0.9% NaCl) Cathode will be placed over the left dorsolateral prefrontal cortex (F3 according to the international EEG system) and anode over the right dorsolateral prefrontal cortex (F4 according to the international EEG system).
  Arms: Cathode tDCS
Device: tDCS Placebo session — This arm will help compare the effects of stimulation versus no stimulation on emotional processing, attentional resources and physiological responses.
  Stimulation will be performed using a tDCS stimulator (Neuroconn or Neuroelectric tDCS stimulator) with two 7×5 cm (35 cm2) sponge electrodes soaked in a saline solution (0.9% NaCl) Anode will be placed over the left dorsolateral prefrontal cortex (F3 according to the international EEG system) and cathode over the right dorsolateral prefrontal cortex (F4 according to the international EEG system)
  Arms: Placebo tDCS

SUMMARY:
The dorsolateral prefrontal cortex (DLPFC) plays a key part in emotional processing and regulation.

Emotions continually influence other cognitive functions such as attentional resources .Emotions also influence a subject's automatic physiological responses .

Transcranial direct current stimulation (tDCS) is an innovative neuro-modulation treatment, often used in major depression.

Various studies have shown that it is possible to modulate emotional processing in healthy subjects, however the impact of this modulation on attentional resources and physiological responses has not been studied. Also, the mechanisms of action of the tDCS on emotional processing are still unclear.

It is necessary to explore the modulation of the DLPFC in healthy subjects in order to better understand the network and mechanisms at stake in the processes.

Thus, investigators plan to study the modulation of the DLPFC (left and right) by tDCS (anode, cathode and placebo) on the processing of emotions and the impact on attentional resources, and physiological responses.

DETAILED DESCRIPTION:
To study the modulation of the DLPFC (left and right) by tDCS (anode, cathode and placebo) on the processing of emotions and the impact on attentional resources, and physiological responses, subjects will undertake 3 tasks before and after a unique tDCS session of 30 minutes.

The first task is a facial expression recognition task, the second measures the attentional processing of emotional information ("Free-viewing task") and the last task focuses on working memory (digit sorting task).

Each task has its cognitive variables but physiological responses will also be measured during each task before and after the tDCS session (Eye movement, i.e. Pupil dilatation and time spent on region of interest; heart rate, skin conductance and respiratory frequency).

3 arms will take part in the study: Anode tDCS Cathode tDCS Placebo tDCS These 3 types of tDCS stimulation will enable us to study the different modulations possible for the DLPFC and the impact on all the variables previously mentioned.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 65 years
* Written given consent

Exclusion Criteria:

* Psychiatric disorder
* Refusal from the subject
* Addiction except for tobacco addiction
* Ocular disease (except from refraction disorders), neurologic or cardiac disease.
* Neuroleptic or anticonvulsivant treatment
* presence of a specific contraindication for tDCS (e.g., personal history of epilepsy, metallic head implant, cardiac pacemaker)
* pregnant or breastfeeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2019-02-12 (Actual); Study Completion 2019-02-12 (Actual)

PRIMARY OUTCOMES:
Performance on a facial expression recognition task | Change from baseline on a facial expression recognition task at one day
  A computerized facial expression recognition task was designed for the study. 240 pictures of emotional faces (8 identities, expressing anger, sadness, happiness, surprise, disgust, or fear, morphed with intensity of 20, 40, 50, 60 and 80%) are randomly displayed on a screen for 500ms. Subjects are asked to identify the emotion by answering on a keyboard.
  Rate of correct responses is the main outcome. During this task, eye movements are recorded by an eye-tracking device. Skin conductance, respiratory and heart rate frequency are also recorded.

SECONDARY OUTCOMES:
Performance on a task measuring the attentional processing of emotional information | baseline
  Computerized "free viewing" attentional task designed for the study. Pairs of emotional faces (neutral/sad ou neutral/happy) are randomly presented on a screen for 3500ms. Subjects are asked to freely explore the faces.
  During this task, eye movements are recorded by an eye-tracking device. Total time spent on Region of Interest (sad, happy or neutral face) is measured.
  Skin conductance, respiratory and heart rate frequency are also recorded.
Performance on a task measuring working memory | baseline
  This working memory task is computerized and designed for this study. It is a digit sorting task in which 5 digits will appear on the screen. After that subjects will mentally have to put the digits in the right order. Subjects will then see a target digit and have to assess whether this target digit is the same as the middle digit in the series previously sorted.
  During this task, pupil dilatation is recorded by an eye-tracking device. Skin conductance, respiratory and heart rate frequency are also recorded.
Eye movements during facial emotion recognition task, attentional task and working memory task | baseline
  total time spent on Region of Interest (for the emotional tasks) and pupil dilatation will be recorded by an SMI RED 250 Eye tracker.
Skin conductance during facial emotion recognition task, attentional task and working memory task | baseline
  this measure will be recorded with a BIOPAC system.
Heart Rate during facial emotion recognition task, attentional task and working memory task | baseline
  this measure will be recorded with a BIOPAC system.
Respiratory frequency during facial emotion recognition task, attentional task and working memory task | baseline
  this measure will be recorded with a BIOPAC system.

CONTACTS AND LOCATIONS:
Overall Officials: HAESEBAERT FREDERIC, PH, Principal Investigator — Vinatier Hospital
Locations (1):
- Ch Le Vinatier, Lyon, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No